CLINICAL TRIAL: NCT06407999
Title: A Prospective, Randomized, Crossover Study on the Effect of Pressure Relief Algorithms (PRA) on Therapy Pressure in APAP Therapy for Obstructive Sleep Apnea (OSA)
Brief Title: Pressure Relief Algorithm Eval
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds were redirected to other projects with higher priority
Sponsor: SleepRes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Home 0002
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will sleep at home with their normal CPAP (continuous positive airway pressure)/APAP (auto-adjusting...) equipment for 4 nights with EPR (expiratory pressure relief) on, the 4 nights with EPR off. The starting therapy will be randomized.
Who Masked: Participant
Masking Description: Participants will not be told which are they are in during any point of the study, although since they are adherent (use their device regularly), they likely will be able to tell.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- APAP w/ EPR On (Experimental): The patient will use their normal CPAP device and equipment in the normal operating mode but we will set EPR on if they do not already use it that way.
  Interventions: Device: Expiratory Pressure Relief
- APAP w/ EPR Off (Placebo Comparator): The patient will use their normal CPAP device and equipment in the normal operating mode but we will set EPR off if they do not already use it that way.
  Interventions: Device: Expiratory Pressure Relief

INTERVENTIONS:
Device: Expiratory Pressure Relief — EPR is a function used in CPAP intended to improve comfort by reducing delivered pressure during the expiratory phase. When EPR is not used, the patient receives true CPAP.
  Other Names: C-Flex, EPR

SUMMARY:
The PRA Effect on APAP Therapy Pressure Study is a randomized, controlled, crossover study in PAP-adherent participants with OSA. Pre-screening is conducted to establish potential eligibility based on regular usage of > 4 hours/night on patients who use an APAP device with a PRA mode. Participants would then be recruited as described below. For those who sign an informed consent, they will be instructed to use the device for the next 8 days with the PRA turned on for four consecutive nights and off for four consecutive nights, but in random orientation. To make sure that the device is not limited to APAP range when adjusting to respond to PRA, the upper limit will be changed to 20 cmH2O during the study. Additionally, only patients who have a current P95 of 8 cmH2O or greater will be eligible so that the maximum PRA setting of 3 cmH2O can be used.

DETAILED DESCRIPTION:
The first phase of recruiting for the PRA Effect on APAP Therapy Pressure Study will be done during a single phone contact following an email recruitment. During this call, participants will be explained the study along with risks and benefits and evaluated for inclusion and exclusion criteria. If the participant is eligible to enter the study, they will be sent an electronic Informed Consent Form to sign. Once the form is signed and verified, the study can then start that evening, after the participant's device has been set for the study.

During both arms of the study, every aspect of operation of the APAP devices will be the same as those the patient normally uses, except for the following three things:

* APAP upper range limit will be set to 20 cmH2O
* PRA or 3 cmH2O will be either on or off
* Participants cannot use a V̇-Com™ device. Participants will randomly be assigned to start with or without PRA. Once the settings are remotely assigned to the device, the patient will sleep on these settings for four nights, ideally consecutively.

After four nights, the PRA setting will be remotely switched to the 2nd arm setting (on or off), and median and P95 pressure, Usage, AHI, and Leak averaged over those four nights will be downloaded. The participant will then use the device with the new settings for an additional four nights, hopefully also sequentially.

Following the 2nd group of four nights, median and P95 pressure, Usage, AHI, and Leak averaged over those four nights will be downloaded, the participant will be informed that their involvement in the study is complete, and the device will be remotely set back to the settings it had prior to the study. Participants will then receive the compensation credit.

ELIGIBILITY:
Inclusion Criteria:

1. Adherent use of ≥ four hours/night over previous 2 months.
2. P95 ≥ 8 cmH2O.

Exclusion Criteria:

1. Excessive alcohol consumption (>14 drinks/week).
2. The use of any illegal drug(s).
3. Any condition that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
P95/P90 | Averaged over every night for each 4-night arm
  P95/P90 represent pressure levels that eliminate breathing obstructions for at least 90% to 95% of the sleep period

SECONDARY OUTCOMES:
Leak | Averaged over every night for each 4-night arm
  Leak measured by the device in excess of the required exhaust valve leak to purge CO2 from the breathing circuit.
Usage | Averaged over every night for each 4-night arm
  Elapsed therapy usage time measured each night
AHI | Averaged over every night for each 4-night arm
  Apnea/Hypopnea Index - Measurement of obstructive events averaged over the night in events per hour.

CONTACTS AND LOCATIONS:
Overall Officials: William H Noah, MD, Study Director — SleepRes, LLC., Sleep Centers of Middle Tennessee, LLC
Locations (1):
- Sleep Centers of Middle Tennessee, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Only plan to publish results.